CLINICAL TRIAL: NCT02434549
Title: Botulinum Toxin-A as a Treatment for Chronic Muscle-Related Pain in Adults With Spastic Cerebral Palsy: a Randomized Controlled Trial
Acronym: BATCP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on efficacy results from interim analysis
Sponsor: Kristina Tedroff (Other)
Collaborators: Danderyd Hospital (Other); Karolinska University Hospital (Other)
Responsible Party: Sponsor-Investigator, Kristina Tedroff, MD, PhD. Associate Professor. Senior Consultant Physician., Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BATCP
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Pain; Cerebral Palsy, Spastic
Keywords: Randomized Controlled Trial; Placebo Controlled; Double Blinded; Botulinum Toxin Type A; Adults; Pain; Spasticity; Cerebral Palsy, Spastic; Dysport
MeSH Terms: conditions — Pain; Cerebral Palsy; Muscle Spasticity | interventions — abobotulinumtoxinA; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botulinum toxin-A (Dysport®) (Active Comparator): Intramuscular injections of Botulinum toxin-A in spastic muscles with regional muscle-related pain
  Interventions: Drug: Dysport®
- Normal saline (Placebo Comparator): Intramuscular injections of normal saline solution in spastic muscles with regional muscle-related pain
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dysport® — Intramuscular injections in spastic muscle with regional muscle-related pain
  Other Names: AbobotulinumtoxinA
  Arms: Botulinum toxin-A (Dysport®)
Drug: Normal saline — Intramuscular injections in spastic muscle with regional muscle-related pain
  Other Names: 0.9 % NaCl; Physiological saline
  Arms: Normal saline

SUMMARY:
The purpose of this double-blinded, placebo-controlled study is to test if treatment with Botulinum toxin-A is effective in reducing chronic muscle-related pain in adults with spastic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Spastic Cerebral Palsy.
* Chronic pain, related to spastic muscle. Chronic pain defined as: 1)Recurring regional pain for at least three months AND 2)Pain intensity on average for the last 24 hours ≥3 on Numerical Rating Scale.
* Signed Informed consent.

Exclusion Criteria:

* Allergy/hypersensitivity to Dysport® or any of its components.
* Pregnancy.
* Women who breastfeed their children.
* Treatment with Botulinum toxin-A within the last five months.
* If there has been dose changes in any muscle-tone altering medication within two weeks of Visit 1.
* A clear degenerative cause behind the pain as elucidated by the clinical examination (e.g. history of osteoarthritis).
* Intellectual disability and/or communication impairment that disable the individual from answering the questionnaires and giving informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-08; Primary Completion 2018-01-26 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Six weeks after treatment
  Proportion of responders derived as reduction of intensity of pain of ≥2 points on the Numerical Rating Scale (NRS) at Visit 3 (six weeks after treatment) compared to baseline.

SECONDARY OUTCOMES:
Use of other analgesic treatment | Six weeks after treatment
  Categories of change in the use of analgesic treatments, derived as Increase, No change, or Decrease at Visit 3 (six weeks after treatment), compared to baseline.
Pain interference | Six weeks after treatment
  Proportion of responders derived as a reduction in mean interference score of ≥1 on the Brief Pain Inventory (BPI-SF) at Visit 3 (six weeks after treatment) compared to baseline.

OTHER OUTCOMES:
HRQoL (Health-Related Quality of Life) | Six weeks after treatment
  Mean change at Visit 3 (six weeks after treatment) compared to baseline in the Short Form 36 v2 Health-related Quality of Life questionnaire (SF-36v2)
Global Impression of Change | Six weeks after treatment
  Proportion of responders at Visit 3 (six weeks after treatment) in the Global Impression of Change Scale (PGIC) derived as at least "Minimally improved".
Fatigue Severity Scale | Six weeks after treatment
  Proportion of responders at Visit 3 (six weeks after treatment) in the Fatigue Severity Scale (FSS) derived as a reduction in mean score of ≥1 point.
Spasticity | Six weeks after treatment
  Proportion of responders at Visit 3 (six weeks after treatment) derived as achieving reduction of spasticity of >1 scale steps on the Modified Ashworth Scale (MAS)
Range of Motion | Six weeks after treatment
  Proportion of responders at Visit 3 (six weeks after treatment) derived as improvement in passive joint range of motion (ROM) ≥ 10 degrees.
Adverse Events | Six weeks after treatment
  Frequency of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Tedroff, MD, PhD, Principal Investigator — Associate Professor, Department of Women's and Children's Health, Karolinska Institutet. Senior Consultant Physician, Astrid Lindgren's Children's Hospital, Stockholm, Sweden.
Locations (2):
- Sweden (2):
  - Department of Rehabilitation Medicine at Danderyd Hospital AB, Danderyd
  - Astrid Lindgren's Children's Hospital at Karolinska University Hospital, Stockholm

REFERENCES:
- [Derived] Jacobson D, Lowing K, Kullander K, Rydh BM, Tedroff K. A First Clinical Trial on Botulinum Toxin-A for Chronic Muscle-Related Pain in Cerebral Palsy. Front Neurol. 2021 Aug 16;12:696218. doi: 10.3389/fneur.2021.696218. eCollection 2021. PMID 34484101